CLINICAL TRIAL: NCT00002580
Title: PROTOCOL FOR THE SCOTTISH PREMENOPAUSAL CHEMO-ENDOCRINE TRIAL
Brief Title: Tamoxifen, Ovarian Ablation, and/or Combination Chemotherapy in Treating Premenopausal Women With Stage I, Stage II, or Stage IIIA Invasive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Scottish Cancer Therapy Network (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063695; SCTN-BR9401; EU-94002; UKCCCR-ABC/BR9401
Record Dates: First submitted 1999-11-01; First posted 2004-03-11 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2007-05

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Fluorouracil; Goserelin; Leuprolide; Methotrexate; Tamoxifen; Laparoscopy; Ovariectomy; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Drug: fluorouracil
Drug: goserelin acetate
Drug: leuprolide acetate
Drug: methotrexate
Drug: tamoxifen citrate
Procedure: conventional surgery
Procedure: laparoscopic surgery
Procedure: oophorectomy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen. Chemotherapy uses different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with hormone therapy may kill more tumor cells. It is not yet known which treatment regimen is most effective for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of tamoxifen with that of ovarian ablation, and/or combination chemotherapy in treating premenopausal women with stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the potential benefits of adjuvant tamoxifen with or without ovarian suppression and/or cyclophosphamide, methotrexate, and fluorouracil (CMF) in premenopausal women with stage I-IIIA, unilateral, invasive breast cancer.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to nodal status (positive vs negative or unknown) and hospital region. Patients undergo surgical resection with or without local radiotherapy, as appropriate. Radiotherapy begins within 8 weeks after surgery for patients randomized to arm I or III and within 4 weeks after completion of chemotherapy for patients randomized to arm II or IV. Patients are randomized to 1 of 4 treatment arms, preferably within 2 weeks after surgery. Arm I: Beginning within 4 weeks after surgery, patients receive oral tamoxifen daily. Treatment continues for 5 years in the absence of disease progression or unacceptable toxicity. Arm II: Beginning within 4 weeks after surgery, patients receive tamoxifen as in arm I and cyclophosphamide IV, methotrexate IV, and fluorouracil IV (CMF) on day 1. Chemotherapy continues every 3 weeks for 6 courses. Arm III: Beginning within 4 weeks after surgery, patients receive tamoxifen as in arm I and 1 of 3 ovarian suppression regimens, preferably regimen A. Regimen B is the preferred alternative to regimen A. Regimen A: Patients undergo oophorectomy. Regimen B: Patients undergo radiation-induced menopause comprising radiotherapy to the pelvis on days 1-4. Regimen C: Beginning 4 weeks after surgery, patients receive goserelin subcutaneously (SC) or leuprolide SC or intramuscularly on day 1. Treatment continues every 4 weeks for 2 years. Arm IV: Patients receive tamoxifen as in arm I and CMF as in arm II followed within 4 weeks by ovarian suppression as in arm III. Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A total of 1,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven unilateral, invasive breast cancer Stage T0-3, N0-1, M0 No carcinoma in situ alone, including Paget's disease of the nipple without underlying invasion No evidence of distant disease, including ipsilateral supraclavicular node enlargement unless proven benign No history of pure carcinoma in situ in either breast Hormone receptor status: Not specified

PATIENT CHARACTERISTICS: Age: 70 and under Sex: Female Menopausal status: Premenopausal, defined by 1 of the following criteria: Last menstrual period less than 1 year before surgery Under age 50 with prior hysterectomy (for nonmalignant reason) without bilateral oophorectomy Under age 50 and on continuous oral contraception If at variance with the above definitions, hormonal assays in the premenopausal range take precedence Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing No other serious illness No other prior invasive malignancy except adequately treated basal cell or squamous cell skin cancer

PRIOR CONCURRENT THERAPY: Not specified

Max Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 1993-06

CONTACTS AND LOCATIONS:
Overall Officials: W.D. George, MD, MS, FRCS, Study Chair — University of Glasgow
Locations (10):
- United Kingdom (10):
  - University Hospitals of Leicester, Leicester, England
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland
  - Beatson Oncology Centre, Glasgow, Scotland
  - University of Glasgow, Glasgow, Scotland
  - Raigmore Hospital, Inverness, Scotland
  - Royal Alexandra Hospital, Paisley, Scotland
  - Ayr Hospital, Ayr
  - Falkirk Royal Infirmary, Falkirk

REFERENCES:
- [Result] Featherstone C, Harnett AN, Brunt AM. Ultrasound localization of the ovaries for radiation-induced ovarian ablation. Clin Oncol (R Coll Radiol). 1999;11(6):393-7. doi: 10.1053/clon.1999.9090. PMID 10663329